CLINICAL TRIAL: NCT07145151
Title: A Phase 2, Randomized, Double-blind, Parallel-group, Placebo-controlled Study to Evaluate the Efficacy and Safety of UBT251 Injection in Adult Patients With Metabolic Dysfunction-associated Steatohepatitis (MASH)
Brief Title: A Study of UBT251 in Participants With Metabolic Dysfunction-Associated Steatohepatitis (MASH)
Acronym: MASH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The United Bio-Technology (Hengqin) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TUL-UBT251（Ⅱ-3）202501; Approved No.:2023LP01795 (Other: National Medical Products Administration)
Record Dates: First submitted 2025-08-13; First posted 2025-08-28 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-08

CONDITIONS: Metabolic Dysfunction-associated Steatohepatitis (MASH)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- UBT251 Low Dose (Experimental): Dose level 1,SC, once a week for 4 weeks; Dose level 2,SC, once a week for 4 weeks; Dose level 3,SC,once a week for 4 weeks; Dose level 3,SC, once a week for 36 weeks.
  Interventions: Drug: UBT251
- Placebo (Placebo Comparator): Placebo administered subcutaneously (SC) once a week for 48 weeks.
  Interventions: Drug: Placebo
- UBT251 Middle Dose (Experimental): Dose level 2,SC, once a week for 4 weeks; Dose level 3,SC, once a week for 4 weeks; Dose level 4,SC,once a week for 4 weeks; Dose level 4,SC, once a week for 36 weeks.
  Interventions: Drug: UBT251
- UBT251 High Dose (Experimental): Dose level 2,SC, once a week for 4 weeks; Dose level 3,SC, once a week for 4 weeks; Dose level 4,SC,once a week for 4 weeks; Dose level 5,SC, once a week for 36 weeks.
  Interventions: Drug: UBT251

INTERVENTIONS:
Drug: UBT251 — UBT251 administered subcutaneously (SC) once a week.
  Arms: UBT251 High Dose; UBT251 Low Dose; UBT251 Middle Dose
Drug: Placebo — Placebo,SC,once a week for 48 weeks
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Phase 2 clinical study evaluating the efficacy and safety of UBT251 in MASH subjects. Subjects will be randomly assigned to UBT251 2mg-dose, 4mg-dose，6mg-dose and placebo groups. The entire trial cycle includes a 6-week screening period, a 48-week double-blind treatment period, and a 4-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

Age 18-75 years (inclusive) at screening; sex unrestricted.

Subjects with centrally confirmed MASH (metabolic dysfunction-associated steatohepatitis) based on liver histopathology must meet all the following criteria:

1. NAS (Appendix 1) ≥ 4 （with at least 1 point each for lobular inflammation and ballooning degeneration）;
2. CRN fibrosis stage (see Appendix 2) of F2 or F3 (a liver biopsy obtained ≤ 6 months before screening is acceptable if it meets the above criteria).

3.Magnetic Resonance Imaging-Proton Density Fat Fraction (MRI-PDFF) ≥ 8 % at screening (MRI-PDFF results obtained within 2 months prior to screening at the trial site are acceptable).

4.Subjects must have <5% body weight fluctuation during the 6 weeks prior to randomization (based on self-reported data), calculated as: [(Highest weight - Lowest weight) / Highest weight] × 100%. For subjects using historical liver biopsy, documented weight change from biopsy to randomization must also be < 5 %.

5.At least one cardiometabolic risk factor at screening:

1. Body mass index (BMI) ≥ 24.0 kg/m², or waist circumference ≥90 cm for males or ≥85 cm for females;
2. Blood pressure ≥ 130/85 mmHg, or on antihypertensive therapy;
3. Fasting triglycerides ≥ 1.70 mmol/L and < 5.6 mmol/L, or on lipid-lowering therapy;
4. Fasting HDL-C ≤ 1.0 mmol/L for males or ≤ 1.3 mmol/L for females; or on lipid-lowering therapy;
5. Fasting glucose ≥ 6.1 mmol/L or glycated hemoglobin (HbA1c) ≥ 5.7 %, or documented history of type 2 diabetes mellitus (T2DM), or Homeostatic Model Assessment of Insulin Resistance index ≥ 2.5.

6.Subjects with type 2 diabetes mellitus (T2DM) must meet glycated hemoglobin (HbA1c) ≤ 9.0 % at screening (local result obtained ≤ 2 weeks before randomization accepted), and stable glycemic control regimen for at least 3 months prior to screening: subjects must be on diet and exercise control alone, or in combination with stable-dose glucose-lowering medications, with the following requirements::

1. Diet and exercise alone;
2. Stable-dose use of metformin, sulfonylureas, sodium-glucose cotransporter-2 (SGLT2) inhibitors, or insulin, stable insulin dose defined as ≤35% variation in total daily insulin dose; 7. Subjects (including partners) must have no pregnancy plans from screening through 6 months post-trial and must practice contraception during the study, with no plans to donate sperm/oocytes for 6 months after trial completion.

8. Subjects must provide informed consent prior to trial participation and voluntarily sign the written informed consent form.

9.Voluntarily comply with all trial follow-up requirements, demonstrate good protocol adherence, and be willing and able to undergo protocol-specified liver biopsies.

Exclusion Criteria:

1. Known hypersensitivity to the investigational product or any of its excipients, or allergy to other GLP-1 receptor agonists, or clinically significant history of multiple/severe drug allergies, or current allergic diseases or hypersensitivity diathesis;
2. Previous use of any of the following drugs or treatments:

1) Use of GLP-1 receptor agonists (GLP-1R), or GLP-1R/GCGR agonists, or GLP-1R/GIPR/GCGR agonists within 3 months prior to screening; 2) Cumulative use for ≥4 weeks within 3 months prior to screening, use within 1 month prior to screening, or planned use during the trial of vitamin E (dose >400 IU/day), thiazolidinediones, polyunsaturated fatty acids, or ursodeoxycholic acid; 3) Cumulative use for ≥4 weeks within 3 months prior to screening, use within 1 month prior to screening, or planned use during the trial of drugs associated with liver injury, hepatic steatosis, or steatohepatitis: including amiodarone, methotrexate, systemic glucocorticoids (dose >5 mg/day prednisone equivalent), estrogens (dose exceeding hormone replacement therapy or contraceptive use), tetracyclines, tamoxifen, anabolic steroids, valproate, or restricted drugs, or any drug deemed likely to interfere with efficacy or safety evaluations; 4) Unstable doses of statins, fibrates, or PCSK9 inhibitors within 1 month prior to screening; 3.History or evidence of any of the following diseases:

1. Chronic liver disease other than MASH (e.g., autoimmune liver disease, primary biliary cholangitis, primary sclerosing cholangitis, chronic liver disease-related ascites, esophageal varices, hepatic encephalopathy, etc.).
2. Diagnosis of type 1 diabetes or other specific types of diabetes, except resolved gestational diabetes;
3. Acute pancreatitis or chronic pancreatitis within 1 year prior to screening, history of pancreatic surgery; or symptomatic gallbladder disease within 1 year prior to screening (e.g., choledocholithiasis, multiple gallstones, etc., except those who underwent cholecystectomy or stone removal);
4. Personal or family history (first-degree relatives-parents, children, or siblings) of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN2);
5. History of severe psychiatric disorders, including but not limited to depression, suicidal tendencies or attempts, schizophrenia, bipolar disorder, etc.;
6. Clinically significant active cardiovascular/cerebrovascular disease within 6 months prior to screening, defined as: ① Myocardial infarction (MI) or unstable angina; ② Cardiac-related surgery (including coronary artery bypass grafting, percutaneous coronary intervention); ③Congestive heart failure (New York Heart Association [NYHA] Class III-IV) (see Appendix 3); ④ Cerebrovascular accident (except old lacunar infarction), including but not limited to stroke/transient ischemic attack; ⑤ Other cardiovascular or cerebrovascular diseases deemed unsuitable for trial participation by the investigator;
7. Retinal diseases requiring urgent treatment at screening (including but not limited to retinal vascular disorders, retinal inflammation, retinal detachment, retinal degeneration, etc.), as assessed by the investigator;
8. History of severe hypoglycemic coma or frequent hypoglycemia (≥1 episode/week) within 2 months prior to enrollment (defined as fingertip or venous blood glucose <3.9 mmol/L for T2DM subjects or <2.8 mmol/L for non-T2DM subjects);
9. Gastroparesis or other gastrointestinal motility disorders (e.g., pyloric obstruction, intestinal obstruction, etc.), uncontrolled gastroesophageal reflux disease, or gastrointestinal conditions deemed by the investigator to increase drug-related risks (e.g., severe active ulcers, inflammatory bowel disease, acute gastroenteritis, symptomatic chronic gastritis, functional gastrointestinal disorders, intestinal tuberculosis, etc.);
10. Major surgery, severe trauma, or severe infection within 1 month prior to screening, deemed unsuitable for participation by the investigator;
11. History of malignancy (except adequately treated cervical carcinoma in situ, basal or squamous cell skin cancer, localized prostate cancer post-radical therapy, ductal carcinoma in situ of the breast post-radical therapy, and papillary thyroid carcinoma post-radical therapy);
12. Concurrent diseases deemed by the investigator to affect subject safety, efficacy evaluation, or compliance, e.g., neurological, endocrine, psychiatric, etc. ; 4.Laboratory abnormalities at screening meeting any of the following criteria:

1) Hepatic or renal impairment, based on each hospital laboratory's reference values, serum ALT and/or AST >5× upper limit of normal (ULN); serum total bilirubin ≥1.5×ULN; estimated glomerular filtration rate (eGFR) <60 mL·min-1·1.73m-2. (calculated using CKD-EPI formula see Appendix 4) ; 2) Alkaline phosphatase (ALP) >2.0×ULN; 3) Platelet count < 100 × 10⁹/L; 4) Serum calcitonin ≥ 50 pg/mL (i.e., 50 ng/L); 5) Serum amylase or lipase > 2.0× ULN; 6) International normalized ratio (INR) >1.2×ULN at screening; 7) Albumin < 3.5 g/dL (35.0 g/L). 8) Uncontrolled hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg at screening), subjects may be re-screened after 1 month of initiating or adjusting antihypertensive therapy; 9) Unstable thyroid dysfunction requiring medication adjustment at screening, or clinically significant abnormal thyroid function test results necessitating treatment initiation; 10) Subjects with clinically significant ECG abnormalities at screening, including: a) Second- or third-degree atrioventricular block; b) Long QT syndrome, QTcF >470 ms for females or >450 ms for males (QTcF = QT/(RR^0.33) ); c) Wolff-Parkinson-White syndrome; or d) Other severe arrhythmias requiring treatment; 11) Abnormal physical examination, vital signs, or laboratory results deemed clinically significant by the investigator, potentially posing major risks or interfering with efficacy, safety, or PK evaluations; 5.Contraindications to liver biopsy at screening, as assessed by the investigator:(1) Hepatic hemangioma or hepatic alveolar echinococcosis;(2) Extrahepatic obstructive jaundice;(3) Significant bleeding tendency, severe thrombocytopenia, or coagulation disorders;(4) Coma or uncooperative due to other conditions;(5) Infection at the puncture site; 6.Positive for hepatitis B surface antigen, positive for hepatitis B core antibody (except those with positive anti-HBc but hepatitis B virus deoxyribonucleic acid [HBV-DNA] below the lower limit of the reference range), positive for hepatitis C virus antibody with hepatitis C virus ribonucleic acid (HCV-RNA) above the upper limit of the reference range (subjects with a history of HCV infection may be enrolled if HCV PCR has been negative for more than 3 years), positive for human immunodeficiency virus antibody, or positive for syphilis antibody (except cured syphilis) will be excluded; 7.Blood loss or donation > 400 mL within 3 months prior to screening, receipt of blood/component transfusions; or concurrent hemoglobinopathy, hemolytic anemia, or sickle-cell disease.

8.MRI contraindications, including but not limited to severe claustrophobia, large tattoos, inner ear implants, pacemakers or other implantable rhythm management devices, MRI-incompatible intracranial aneurysm clips, or other non-MRI-compatible metal implants (e.g., insulin pumps, hip replacements); 9.Participation in other clinical trial within 3 months prior to screening or 5 half-lives of the investigational drug (whichever is longer)(except for screening-only or non-interventional studies): 10.Excessive alcohol consumption within 12 months prior to screening, defined as >210 g/week (male) or >140 g/week (female) of ethanol (alcohol) for >3 months. Ethanol intake [g] = volume [mL] × alcohol percentage × 0.8); 11.Lactating or pregnant females; 12.Intolerance to venipuncture or history of needle/phobia; 13.Other conditions deemed unsuitable for trial participation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2027-06-04 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With MASH resolution With no Worsening of Fibrosis on Liver Histology | Baseline, Week 48

SECONDARY OUTCOMES:
Proportion of Participants with MASH improvement with a ≥1-stage histological improvement in liver fibrosis. | Baseline, Week 48
Proportion of Participants with MASH resolution with a ≥1-stage histological improvement in liver fibrosis. | Baseline, Week 48
Percentage of Participants With ≥1 Point Decrease in Fibrosis Stage With No Worsening of MASH on Liver Histology | Baseline, Week 48
Mean Absolute Change and Percent Change from Baseline in Body Weight [kg] | Baseline, Week 12, Week 24, Week 48
Changes from baseline in waist circumference[cm] | Baseline, Week 12, Week 24, Week 48
Changes from baseline in waist-to-hip ratio[%] | Baseline, Week 12, Week 24, Week 48
Change from baseline in liver stiffness measurement (LSM) and controlled attenuation parameter (CAP). | Baseline, Week 24, Week 48
Percentage change from baseline in MRI-PDFF. | Baseline, Week 24, Week 48
Proportion of subjects achieving >30%, >50%, or >70% reduction in MRI-PDFF from baseline. | Baseline, Week 24, Week 48
Mean Absolute Change and Percentage change From Baseline in triglyceride [mmol/L] | Baseline, Week 12, Week 24, Week 48
Mean Absolute Change and Percentage change From Baseline in total cholesterol[mmol/L] | Baseline, Week 12, Week 24, Week 48
Mean Absolute Change and Percentage change From Baseline in low-density lipoprotein cholesterol[mmol/L] | Baseline, Week 12, Week 24, Week 48
Mean Absolute Change and Percentage change From Baseline in high-density lipoprotein cholesterol[mmol/L] | Baseline, Week 12, Week 24, Week 48
Changes from baseline in fasting insulin (FINS) | Baseline, Week 24, Week 48
Change from Baseline in homeostatic model assessment of insulin resistance (HOMA-IR) | Baseline, Week 24, Week 48
Change from Baseline in Homeostasis Model Assessment of β-cell function (HOMA-β) | Baseline, Week 24, Week 48
Percentage change from baseline in hepatic enzymes alanine aminotransferase (ALT) [%] | Baseline, Week 12, Week 24, Week 48
Percentage change from baseline in hepatic enzymes aspartate aminotransferase (AST) [%] | Baseline, Week 12, Week 24, Week 48
Percentage change from baseline in cytokeratin-18 (CK18) fragments[%] | Baseline, Week 12, Week 24, Week 48
Percentage change from baseline in type III procollagen N-terminal propeptide (Pro-C3)[%] | Baseline, Week 12, Week 24, Week 48
Percentage change from baseline in high-sensitivity C-reactive protein (hsCRP)[%] | Baseline, Week 12, Week 24, Week 48
Change from baseline in scores in Fibrosis-4 Index (FIB-4) | Baseline, Week 12, Week 24, Week 48
Change from baseline in scores in Enhanced Liver Fibrosis (ELF) | Baseline, Week 12, Week 24, Week 48
Change from baseline in scores in NAFLD Fibrosis Score (NFS) | Baseline, Week 12, Week 24, Week 48
Change from baseline in scores in AST-to-Platelet Ratio Index (APRI) | Baseline, Week 12, Week 24, Week 48

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua ChangGung Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No